CLINICAL TRIAL: NCT06659770
Title: A Real-World Observational Study: Zevorcabtagene Autoleucel Injection in Patients with Relapsed/Refractory Multiple Myeloma
Status: Not yet recruiting | Type: Observational
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CT053-MM-05
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-07

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Zevorcabtagene Autoleucel — Zevorcabtagene Autoleucel is a novel fully human BCMA-targeting CAR-T therapy

SUMMARY:
This study is a single-arm, open-label, multicenter, post-marketing, Phase IV, prospective, observational clinical trial to evaluate the efficacy and safety of the post-marketing product zevor-cel as treatment for subjects with R/R MM in the real world.

DETAILED DESCRIPTION:
Primary study endpoints:

Overall Survival Rate (OS Rate) at 24 months after infusion：Survival rate from the start of cell infusion to 24 months after infusion.

Secondary study endpoints:

Incidence and Severity of Treatment-Related Adverse Events (TEAEs) for zevor-cel Incidence and severity of adverse events (AEs) related to study treatment Incidence of serious adverse events (SAEs) related to study treatment

Other efficacy endpoints of zevor-cel:

Overall response rate (ORR)：Proportion of subjects with a partial response (PR) or above.

Complete response or stringent complete response rate (CR/sCR) ：The proportion of subjects with the best response of CR/sCR.

Duration of Response (DOR)：The time from first response to disease progression or death caused by any reasons in subjects with the best response of PR and above.

Progression Free Survival (PFS) Overall survival (OS)： The time from the start of cell infusion to death due to any cause.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Subjects with refractory/relapsed multiple myeloma who meet product indication criteria and have received commercialized zevor-cel infusion.
3. Voluntary participation in this study and willingness to sign the informed consent form, for subjects incapable to provide consent, informed consent must be obtained from their legally acceptable guardians.

Exclusion Criteria:

1. There were no specific exclusion criteria for this study。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted in a medical institution that has been commercially evaluated and certified. Before carrying out the corresponding procedures for the study, the informed consent signed by the subjects themselves must be obtained, and for patients who do not have full civil capacity, the informed consent of their guardians must be obtained.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate long-term survival benefits of zevor-cel in subjects with R/R MM | 24 months
  Statistical analysis of OS will be performed, survival curves of OS will be plotted, and 1-year and 2-year survival rates will be calculated. The median, 25% quantile, and 75% quantile of OS will be calculated with their 95% confidence intervals.

IPD SHARING:
Plan to Share IPD: No